CLINICAL TRIAL: NCT02145442
Title: Effects and Safety of Obex in Overweight and Obese Subjects With or Without Impaired Fasting Glucose
Brief Title: Effects of Obex in Overweight and Obese Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBEX-IFG-2014
Record Dates: First submitted 2014-05-20; First posted 2014-05-23 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Overweight; Obesity
Keywords: Impaired fasting glucose; Prediabetes; Obesity; Overweight; Insulin sensitivity; Weight loss; Nutritional supplement; Waist; Body composition
MeSH Terms: conditions — Overweight; Obesity; Prediabetic State; Insulin Resistance; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Obex (Experimental): Obex®, two oral sachets daily during three months.
  Interventions: Dietary Supplement: Obex

INTERVENTIONS:
Dietary Supplement: Obex — Obex® will be administered two sachets daily dissolved in a glass of water, 30 minutes before lunch and dinner during three months. Participants will be not trained about changes of lifestyle on their diets, or physical activity.

SUMMARY:
* Obesity is an important and growing public health worldwide
* Obesity is highly related to the development of metabolic syndrome, diabetes, cardiovascular diseases and cancer
* An extensive body of evidence from efficacy trials has shown that weight loss is achievable, however, a modest weight loss is achieved in a small proportion of patients
* Important adverse events have been reported with the use of antiobesity drugs.
* The use of natural products with potential effects inducing weight loss is an alternative strategy for treating patients with overweight and obesity. However, efficacy and safety should be evaluated in RCT.
* Obex combines different molecules with potential effects inducing weight loss and control on metabolic parameters such as fasting glucose, cholesterol and triglycerides.
* Therefore, the administration of Obex in overweight and obese patients with impaired fasting glucose could be an excellent strategy to induce weight loss and ameliorate the metabolic disturbances related to obesity and overweight.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and Obese subjects with and without IFG
* Ability to provide informed consent

Exclusion Criteria:

* Presence of diabetes mellitus, hepatic, renal or cardiovascular disease
* Other diseases associated with insulin resistance (eg. Acromegalia, endogenous hypercortisolism, etc)
* Sepsis or any other condition that could potentially interfere with treatment
* History of bariatric surgery
* Pregnancy or lactation
* Concomitant disease with reduced life expectancy
* Severe psychiatric conditions
* Anyone with chronic medical conditions requiring regular intake of any prescription medications.
* Used drugs for weight loss (e.g., Xenical [orlistat], Meridia [sibutramine], Acutrim [phenylpropanolamine], Accomplia [rimonabant], Alli [low-dose orlistat], or other similar over-the-counter weight loss remedies or medications) within 3 months of screening
* Are actively participating in, or have participated in a formal weight loss program within the last 3 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Obex® on fasting glucose levels | Three months of treatment
  The primary outcome is to evaluate the effect of the treatment with Obex® on fasting glucose levels
To determine the safety of serious supplement-related adverse events | Three months of treatment
  Adverse events will be evaluated during the three months of treatment

SECONDARY OUTCOMES:
To evaluate the effect of Obex® on fasting insulin levels | Three months of treatment
  The insulin levels will be evaluated at baseline and at the end of treatment.
• To evaluate the effect of Obex® on insulin sensitivity by homeostasis model assessment-estimated insulin resistance (HOMA-IR), calculated from individual serum measures (fasting insulin x fasting glucose/22.5) | Three months of treatment
  The HOMA-IR will be evaluated at baseline and at the end of treatment.
To evaluate the effect of Obex® on insulin sensitivity by quantitative insulin sensitivity check index, Bennett and Raynaud insulin sensitivity indexes | Three months of treatment
  The Quicki, Bennett and Raynaud insulin sensitivity indexes will be evaluated at baseline and at the end of treatment.
  QUICKI = [1/[log I0 + log G0], Bennett index (BEN) = 1/(log I0 x log G0), Raynaud index (RAY) = [40/I0])
• To evaluate the effect of Obex® on β-cell function by homeostatic model assessment-beta cell (HOMA-β), calculated from individual serum measures (20 x fasting insulin (µU/mL)/fasting glucose (mmol/L)-3.5) | Three months of treatment
  The HOMA-B will be evaluated at baseline and at the end of treatment
• To evaluate the effect of Obex® on cholesterol, triglyceride and high density lipoprotein cholesterol levels (HDL-c) | Three months of treatment
  The cholesterol, triglyceride and HDL-c levels will be evaluated at baseline and at the end of treatment.
To evaluate the effect of Obex® on Glycosylated Hemoglobin (HbA1c) | Three months of treatment
  The HbA1c will be evaluated at baseline and at the end of treatment.
To evaluate the effect of Obex® on the body weight. | Three months of treatment
  The body weight will be measured at baseline and at the end of treatment.
• To evaluate the effect of Obex® on Body Mass Index (BMI) and Conicity Index (CI) | Three months of treatment
  The BMI and CI will be measured at baseline and at the end of treatment.
To evaluate the effect of Obex® on the waist and hip circumferences | Three months of treatment
  Waist and Hip circumferences will be measured at baseline and at the end of treatment.
To evaluate the effect of Obex® on arterial blood pressures (BP) | Three months of treatment
  The arterial BP will be evaluated at baseline and at the end of treatment.
• To evaluate the effect of Obex® on hepatic enzymes (Alanine aminotransferase, Aspartate aminotransferase, gamma-glutamyltransferase, Alkaline Phosphatase) | Three months of treatment
  The hepatic enzymes will be evaluated at baseline and at the end of treatment.
To evaluate the effect of Obex® on creatinine and uric acid concentrations | Three months of treatment
  The creatinine and uric acid levels will be evaluated at baseline and at the end of treatment.
To evaluate the effect of Obex® on haemoglobin and serum iron levels | Three months of treatment
  The haemoglobin and iron levels will be evaluated at baseline and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cabrera, M.D., Ph.D., Principal Investigator — National Institute of Endocrinology, Havana, Cuba
Locations (1):
- National Institute of Endocrinology, Plaza de la Revolución, La Habana, Cuba